CLINICAL TRIAL: NCT01172769
Title: A Single Arm, Open-label Multicenter Phase II Trial of Temsirolimus in Patients With Relapsed/Recurrent Squamous Cell Cancer of the Head and Neck (HNSCC)
Brief Title: Efficacy Study of Temsirolimus to Treat Head and Neck Cancer
Acronym: TEMHEAD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hannover Medical School (Other)
Responsible Party: Principal Investigator, Viktor Grünwald, Associate Professor MD, Hannover Medical School
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HN001
Record Dates: First submitted 2010-07-07; First posted 2010-07-30 (Estimated); Last update posted 2013-11-08 (Estimated); Status verified 2013-11

CONDITIONS: Head and Neck Squamous Cell Carcinoma
Keywords: HNSCC
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — temsirolimus; Sirolimus; Protein Kinase Inhibitors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Temsirolimus (Experimental)
  Interventions: Biological: Temsirolimus

INTERVENTIONS:
Biological: Temsirolimus — After dissolving and dilution 25 mg of temsirolimus will be administered i.v. once a week by 30 minute infusion.
  Study treatment will continue until tumor progression or unless unacceptable toxicity is encountered.
  Other Names: Torisel; mTOR inhibitor; protein kinase inhibitor

SUMMARY:
The purpose of this study is to determine whether temsirolimus is effective in the treatment of relapsed/recurrent squamous cell cancer of the head and neck (HNSCC)

DETAILED DESCRIPTION:
Temsirolimus is an inhibitor of the mammalian target of rapamycin (mTOR), a crucial regulator of cell cycle progression. It was approved in the treatment of advanced renal cell carcinoma. Temsirolimus demonstrated also antitumor activity in a variety of other human cancer models, such as gliomas, rhabdomyosarcomas, neuroblastomas, prostata and breast cancer through induction of apoptosis or inhibition of proliferation. A similar effect was noted in HNSCC cell lines.

This is the first study evaluating the efficacy and safety of temsirolimus in platinum/cetuximab-refractory HNSCC.

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent must be given prior to study inclusion
* Histological or cytological confirmed recurrent or metastatic squamous cell carcinoma of the head and neck (HNSCC)
* Measurable progressive disease after platinum-based radiochemotherapy or recurrence or metastatic progressive disease after 1st line platinum-based chemotherapy
* Patients with loco-regional recurrence need to be progression free for at least 6 months after platinum-based radiochemotherapy, if locoregional recurrence is the only lesion
* Cetuximab must have been included in at least one prior line of therapy
* Disease is not amenable to surgery, radiotherapy or platinum-based chemotherapy
* At least one measurable lesion according to RECIST (Version 1.0) criteria
* Age > 18 years
* ECOG performance status 0-2
* Brain metastases require completion of local therapy with discontinuation of steroids prior to start of treatment
* If of childbearing potential, willingness to use effective contraceptive method (double barrier method) for the study duration and 2 months after last dose
* Willingness and ability to comply with the protocol
* Adequate bone marrow function, liver and renal function

Exclusion Criteria:

* Live expectancy less than 3 months
* Anticancer treatment during the last 30 days prior to start of treatment, including systemic therapy, radiotherapy or major surgery
* Participation in a clinical trial within the last 30 days prior to study treatment
* Serious illness or medical condition other than the disease under study
* Other malignancies within 3 years, with exception of HNSCC, history of a previous basal cell carcinoma of the skin or pre-invasive carcinoma of the cervix
* Inability to potentially complete follow up and treatment per protocol for psychological, familial, sociological or geographical reasons
* Pregnancy or breast feeding
* Known allergic/hypersensitivity reaction to any component of the treatment
* Concurrent treatment with oral anticoagulants
* Uncontrolled diabetes: fasting serum glucose > 2.0 ULN
* Active or uncontrolled infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2010-06; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Progression free rate | at week 12
  The primary endpoint is the patients free of progression (PFR) at week 12 based on CT or MRI scans evaluated according to RECIST criteria.

SECONDARY OUTCOMES:
Time to disease progression | 6 weeks (average)
  time to disease progression
Toxicity of temsirolimus | 12 weeks
  toxicity of temsirolimus are to be evaluated by CTC 3.0 criteria
Objective response rate | at week 12
  objective response rate by RECIST
Overall survival | at week 12
  overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Viktor Gruenwald, MD, Principal Investigator — Medical School Hannover
Locations (7):
- Germany (7):
  - Charitè Berlin Campus Benjamin Franklin Medical Clinic III, Berlin
  - Ev. Bethesda- Johanniter Klinikum GmbH Clinic for Heamatology and medical Oncology, Duisburg
  - Universitaetsklinikum Essen Clinic and Policlinic for internal medicine (Cancerresearch), Essen
  - Universitätsklinikum Halle Clinic and Policlinic of internal Medicine IV, Halle
  - Medical School Hannover Clinic for Heamatology, Hemostaseology, Oncology and stem cell transplantation, Hanover
  - Universitätsklinikum Jena Clinic for Ear, Nose and Throat, Jena
  - Universitätsklinikum Leipzig Clinic and Policlinic for Ear, Nose and Thorat, Leipzig

REFERENCES:
- [Derived] Grunwald V, Keilholz U, Boehm A, Guntinas-Lichius O, Hennemann B, Schmoll HJ, Ivanyi P, Abbas M, Lehmann U, Koch A, Karch A, Zorner A, Gauler TC. TEMHEAD: a single-arm multicentre phase II study of temsirolimus in platin- and cetuximab refractory recurrent and/or metastatic squamous cell carcinoma of the head and neck (SCCHN) of the German SCCHN Group (AIO). Ann Oncol. 2015 Mar;26(3):561-7. doi: 10.1093/annonc/mdu571. Epub 2014 Dec 19. PMID 25527417